CLINICAL TRIAL: NCT06865469
Title: Comparing Efficacy of Intravenous Dexmedetomidine and Lidocaine on Postoperative Analgesia in Patients Undergoing Fracture Hip Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hisham Mamdouh Kotp Mohamed, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dex vs lidocaine fracture hip
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Fracture Hip Surgery
MeSH Terms: interventions — Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D (Active Comparator): patients will recive dexmedetomidine i.v. infusion at 0.4 μg/kg/h
  Interventions: Drug: Dexmedetomidine
- Group L (Active Comparator): patients will received 1.5 mg/kg/h lidocaine hydrochloride 2% (400 mg/20 mL) by i.v. infusion.
  Interventions: Drug: Lidocaine Hydrochloride 2%

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine will be administered by i.v. infusion at 0.4 μg/kg/h
  Arms: Group D
Drug: Lidocaine Hydrochloride 2% — lidocaine hydrochloride 2% (400 mg/20 mL) 1.5 mg/kg/h by i.v. infusion.
  Arms: Group L

SUMMARY:
Perioperative pain management has been a major challenge for anesthesiologists, and there have been persistent efforts to bring out the best possible analgesic technique with the least side effects.

Hip fractures are devastating injuries, constituting a global public health burden and remain one of the largest healthcare challenges of the 21st century. The incidence increases with advancing age and the number of hip fractures is expected to increase to 6.26 million per year in 2050.

Hip fractures impact on patient's psychological, functional, and social wellbeing, and account for substantial healthcare system costs.

Drugs of potential interest such as intravenous (i.v.) lidocaine and dexmedetomidine have been administered both intra and/or postoperatively to decrease perioperative pain and improve other outcomes. Lidoocaine has analgesic, anti inflammatory, and anti hyperalgesia properties.

Several studies have demonstrated that perioperative lidocaine infusion reduces postoperative pain intensity and opioid consumption .

Ease of availability, cost effectiveness, simplicity of administration, safety, and analgesic action make lignocaine an attractive option.

Dexmedetomidine is a highly selective and specific α2 adrenoceptor agonist with useful analgesic, sedative, anxiolytic, and sympatholytic properties.

I.V. dexmedetomidine has gained immense popularity owing to its efficacy as an analgesic adjuvant, translating into reduced opioid consumption.

Intraoperative dexmedetomidine and lignocaine also confirm the enhanced recovery after surgery protocol advocating the reduction of opioid use.

While numerous studies have analyzed i.v. lidoocaine and dexmedetomidine versus placebo regarding postoperative analgesia and outcomes, researches and evidence in the context of minimally invasive surgeries regarding adverse effect profile, postoperative analgesic requirement, perioperative analgesia, anesthesia recovery, and opioid requirements are always welcome(rephrase). Our study was conducted to analyze the effects of intraoperative i.v. lidocaine and dexmedetomidine on pain relief, intra- and postoperative opioid consumption, and effects of these infusions on intraoperative hemodynamic parameters and to evaluate the side effect profiles the aim of the study to analyze the effects of intraoperative intravenous lignocaine/dexmedetomidine on postoperative pain relief and analgesit consumption

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* patients with both sex
* patients who are American society of Anesthesiologists class I or II

Exclusion Criteria:

refusal.

* body mass index (BMI) ≥40 kg/m2.
* History of hypersensitivity to the drugs being evaluated
* Inability to comprehend postoperatively the pain assessment scale/neuropsychiatric disorders.
* chronic use of opioids and opioid addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
pain score NRS score | 24 hours
  The severity of pain will be assessed postoperatively using a 10 cm NRS (0 = no pain and 10 = worst imaginable pain) at rest and coughing at 0, 2nd, 4th, 6th, 12th, 18th, and 24th hours